CLINICAL TRIAL: NCT03299062
Title: Smell, Voice and Nasal Swabs as Markers for Neuro-degenerative Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 206829
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer Disease; Neurodegenerative Diseases
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases | interventions — Cytological Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Parkinson's Disease with Voice Dysfunction Patients (Active Comparator): • Twenty people with Parkinson's Disease requiring evaluation of voice dysfunction by an Ear, Nose, and Throat (ENT) doctor
  Interventions: Diagnostic Test: Cytology and Immunohistochemistry
- Other Neurodegenerative Disorders with Voice Dysfunction (Active Comparator): • Twenty people with other neurodegenerative disorders requiring evaluation of voice dysfunction by an ENT doctor.
  Interventions: Diagnostic Test: Cytology and Immunohistochemistry
- Voice Dysfunction (Placebo Comparator): Twenty people with voice tremor and/or presbylarynx, but no evidence of Parkinson's other neurodegenerative disease, requiring evaluation of voice dysfunction by an ENT doctor.
  Interventions: Diagnostic Test: Cytology and Immunohistochemistry

INTERVENTIONS:
Diagnostic Test: Cytology and Immunohistochemistry — Determine if nasal swabs can provide an adequate sample for evaluation using cytology and immunohistochemistry for alpha-synuclein, A-beta and p-tau staining.

SUMMARY:
Degenerative dementias including Alzheimer's Disease (AD), Parkinson's Disease with Dementia (PDD), Dementia with Lewy Bodies (DLB), Frontotemporal Dementias (FTLD), Corticobasal Degeneration (CBD) and Progressive Supranuclear Palsy (PSP) constitute a significant, and growing burden with an estimated cost to the US healthcare system for 2016 of $236 Billion (1). Definitive diagnosis of these dementias is based on pathological criterion upon autopsy, which presents a significant challenge to establish diagnosis in living patients. Although clinical diagnostic criteria have been developed for several of these disorders, including for Alzheimer's Disease (AD) by the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimers Disease and Related Disorders Association (NINCDS-ADRDA) , Parkinson's Disease (PD) by the United Kingdom Parkinson Disease Brain Bank Diagnostic Criteria (UKPDBB) diagnostic criteria for Parkinson Disease(4) and others, the currently available tests, including the use of imaging markers and Cerebrospinal Fluid (CSF) biological markers do not provide a definite diagnosis since this requires the observation of characteristic neuropathological changes in specific regions of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease, progressive supranuclear palsy, Alzheimer's disease or Mild Cognitive Impairment based on consensus criteria, or suspicion of presbylarynx based on clinical evaluation.
* Require evaluation of voice dysfunction by an ENT doctor given symptoms of impaired voice volume or quality
* Age ≥ 18 years-old to ≤ 90-years old.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active nose bleeds, or abnormal anatomy of the nose that prevent safe nasal swabs, or active oropharyngeal disease that prevents laryngoscopy or voice assessments.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Dhall, MD, MSPH, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parkinson's Disease With Voice Dysfunction Patients | Other Neurodegenerative Disorders With Voice Dysfunction
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment was stopped due to COVID-19 pandemic after 4 subjects with PD and 5 with other neurodegenerative disorders with voice dysfunction were enrolled.
Groups:
- Parkinson's Disease With Voice Dysfunction Patients: • Enrollment was stopped due to COVID-19 pandemic after 4 people with Parkinson's Disease requiring evaluation of voice dysfunction by an Ear, Nose, and Throat (ENT) doctor were enrolled.
  Cytology and Immunohistochemistry: Samples from 1 subject were processed for GFAP and S100 staining to confirm presence of olfactory neuronal tissue.
- Other Neurodegenerative Disorders With Voice Dysfunction: • Enrollment was stopped due to COVID-19 pandemic after 5 people with other neurodegenerative disorders requiring evaluation of voice dysfunction by an ENT doctor.
  Cytology and Immunohistochemistry: No samples were processed for this group.
- Voice Dysfunction: No subjects were enrolled in this arm.
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease With Voice Dysfunction Patients | Other Neurodegenerative Disorders With Voice Dysfunction | Voice Dysfunction | Total
Number analyzed (Participants) | 4 | 5 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 0 | 3
  >=65 years | 4 | 2 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 |  | 4
  Male | 2 | 3 |  | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 5 | 0 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Alpha-synuclein Levels From Nasal Swabs
Description: Determine if nasal swabs can provide an adequate sample for evaluation using cytology and immunohistochemistry for alpha-synuclein, Amyloid-beta (A-beta) and Phospho-tau (p-tau) staining.
Time Frame: Up to 4 weeks after swab is completed
Population: Due to early termination of subject enrollment, there were an insufficient number of samples to process for this analysis. As such, none of the samples were (or will be) analyzed for the outcome measures listed and therefore there are no results to report beyond participant flow.
Groups:
- Parkinson's Disease With Voice Dysfunction Patients: • Enrollment was stopped due to COVID-19 pandemic after 4 people with Parkinson's Disease requiring evaluation of voice dysfunction by an Ear, Nose, and Throat (ENT) doctor were enrolled.
  Cytology and Immunohistochemistry: Although samples from 1 subject were processed for GFAP and S100 staining to confirm presence of olfactory neuronal tissue, none of the samples were (or will be) analyzed for the outcome measures listed and therefore there are no results to report beyond participant flow.
Arm/Group | Parkinson's Disease With Voice Dysfunction Patients | Other Neurodegenerative Disorders With Voice Dysfunction
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was done in a single session for each participant, typically taking 4 hours.
Groups:
- Parkinson's Disease With Voice Dysfunction Patients: Subjects with Parkinson's Disease with Voice Dysfunction Patients
- Other Neurodegenerative Disorders With Voice Dysfunction: Subjects with other Neurodegenerative Disorders with Voice Dysfunction
Arm/Group | Parkinson's Disease With Voice Dysfunction Patients | Other Neurodegenerative Disorders With Voice Dysfunction
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Due to lack of enrollment, and the COVID-19 pandemic, the analysis of biospecimens was not performed. None of the collected samples from this study were analyzed for the outcome measures in this record, and therefore there are no results to report beyond participant flow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03299062/Prot_002.pdf
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03299062/ICF_001.pdf